CLINICAL TRIAL: NCT01018264
Title: URGE-PD: A Multi-site, Double-blind, Randomized, Placebo Controlled Trial of Solifenacin Succinate (VESIcare) for the Treatment of Overactive Bladder in Parkinson's Disease
Brief Title: Solifenacin Succinate (VESIcare) for the Treatment of Overactive Bladder in Parkinson's Disease
Acronym: URGE-PD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Theresa Zesiewicz, MD, Professor of Neurology, University of South Florida
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: URGE-PD
Record Dates: First submitted 2009-11-19; First posted 2009-11-23 (Estimated); Results first posted 2015-05-27 (Estimated); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Overactive Bladder in Parkinson's Disease
Keywords: Overactive bladder; Urinary incontinence; Urinary frequency; Parkinson's disease
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence; Parkinson Disease | interventions — Solifenacin Succinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- solifenacin succinate (VESIcare) (Experimental)
  Interventions: Drug: solifenacin succinate (VESIcare)
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: solifenacin succinate (VESIcare) — up to 10mg every day orally
  Arms: solifenacin succinate (VESIcare)
Drug: placebo — placebo matching solifenacin succinate (VESIcare) up to 10mg orally every day
  Arms: placebo

SUMMARY:
This study will assess the effectiveness of solifenacin succinate (VESIcare) in reducing symptoms of overactive bladder in Parkinson's disease (PD) patients.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients with idiopathic PD according to the UK Parkinson's Disease Society Brain Bank Clinical Diagnosis Criteria.
2. Age 40 years to 80 years.
3. Stable dose of antiparkinsonian medication 4 weeks prior to study entry.
4. Patients must score 1.0 to 3.0 on the Modified Hoehn and Yahr scale.
5. Women of child-bearing potential must use a reliable method of contraception.
6. Must be experiencing symptoms of overactive bladder according to the ICS definition of a minimum voiding 8 or more times/24 hours and a daily average of at least 1 episode of urgency and/or urinary incontinence (urge incontinence predominately as measured by 3IQ diary) per 24 hours during a 3-day micturition diary period. Patients must have documentation of OAB within the last 6 months.
7. The patient must have evidence of PSA less than or equal to 4 (males only) within the last 12 months (obtained from primary care physician).
8. The patient must have had a bladder scan within six months of the screening visit. This scan uses ultrasound technology to measure residual fluid levels in the bladder after urination. This scan must document post void residual of 200 mls or less. A bladder scan printout or a note documenting these findings must be provided before baseline.
9. Clearance from the patient's internist or primary care health provider who has examined the patient within the last 6 months.

Exclusion Criteria:

1. Any illness that in the investigator's opinion preclude participation in this study.
2. Pregnancy or lactation.
3. Concurrent participation in another clinical study.
4. Dementia or other psychiatric illness that prevents the patient from giving informed consent (Mini Mental Status Exam scores less than 27).
5. Legal incapacity or limited legal capacity.
6. History of prostate cancer or Transurethral resection of the prostate (TURP) (males only).
7. Presence of severe renal disease. BUN 50% greater than normal (normal BUN levels should be within a range of 5 to 20 mg/ d L and creatinine between .7 and 1.4 mg/ d L). Labs within the past 12 months will be requested from the patient's health care provider or urologist. If labs are not available within this time-frame or if results are abnormal, labs will be obtained as part of the screening visit.
8. Presence of major hepatic impairment (cirrhosis, viral hepatitis, nonalcoholic steatohepatitis, Wilson's disease, or Hemochromotosis).
9. Currently taking ketaconazole (anti-fungal) or any CYP3A4 inhibitor such as itraconazole, ritonavir, nelfinavir, clarithromycin, or nefazadone.
10. Any history of bladder outflow obstruction or gastrointestinal obstructive disorders.
11. History of narrow angle glaucoma.
12. Patients who have undergone pelvic radiation at any time.
13. Currently taking any of the following medications:

    * Antiarrhythmics: flecainide (Almarytm, Apocard, Ecrinal, Flécaine), digoxin (Lanoxin, Digitek, Lanoxicaps)
    * Antipsychotics: thioridazine (Mellaril, Novorizadine, Thioril)
    * Tricyclic anti-depressants: amitriptyline (Elavil, Tryptanol, Endep, Elatrol, Tryptizol, Trepiline, Laroxyl), amoxapine (Asendin, Asendis, Defanyl, Demolox, Moxadil), clomipramine (Anafranil), desipramine (Norpramin, Pertofrane), imipramine (Antideprin, Deprenil, Deprimin, Deprinol, Depsonil, Dynaprin, Eupramin, Imipramil, Irmin, Janimine, Melipramin, Surplix, Tofranil), nortriptyline (Aventyl, Pamelor, Nortrilen), protriptyline (Vivactil), trimipramine (Stangyl, Surmontil, Rhotrimine)
    * Psychotropics: doxepin (Aponal, Adapine, Sinquan, Sinequan)
    * Anticholinergics/Antispasmodics: trihexyphenidyl (Artane, Aparkan), benztropine (Cogentin), oxybutynin (Ditropan, Ditropan XL, Lyrinel XL, Oxytrol), darifenacin (Enablex), emepronium, flavoxate (Urispas), meladrazine, propiverine, solifenacin (Vesicare), tolterodine (Detrol, Detrol LA), trospium (Sanctura)
    * Selective Serotonin-Norepinephrine Reuptake Inhibitors (SNRI): duloxetine (Cymbalta, Yentreve), Venlafaxine (Effexor, Effexor XR)
    * Arylalkylamines: pseudoephedrine (Sudafed)
    * Anti-androgen: bicalutamide (Casodex, Cosudex, Calutide, Kalumid), finasteride (Proscar, Propecia, Fincar, Finpecia, Finax, Finast, Finara, Finalo, Prosteride, Gefina, Finasterid IVAX), dutasteride (Avodart, Avidart, Avolve, Duagen, Dutas, Dutagen, Duprost), Zoladex (goserelin acetate), Eulexin (flutamide), Lupron (leuprolide acetate)
    * Antihypertensives: prazosin (Minipress, Vasoflex, Hypovase)
    * Estrogens (Menest, Premarin, Premarin IV)
    * Acetylcholinesterase inhibitors (rivastigmine (Exelon), galantamine, (Reminyl, donepezil (Aricept), Tacrine.
    * Memantine (Namenda)
14. Urinary obstruction in male PD patients as diagnosed by a urologist
15. Active urinary tract infection.
16. Patients with a history of chronic severe constipation (by self report)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Zesiewicz, MD, Principal Investigator — University of South Florida
Locations (3):
- United States (3):
  - University of Miami, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Solifenacin Succinate (VESIcare) | Placebo
Started | 10 | 13
Completed | 9 | 12
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Solifenacin Succinate (VESIcare) | Placebo | Total
Number analyzed (Participants) | 10 | 13 | 23
Age, Customized [Mean (Standard Deviation); unit: years]
  Age (years) | 67.6 (6.6) | 66.5 (9.3) | 66.96 (8.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 7 | 8 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 9 | 12 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 1 | 2
  White | 8 | 10 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Unified Parkinson's Disease Rating Scale (UPDRS) ADL subsection (mean) [Mean (Standard Deviation); unit: units on a scale] — This subscale of the UPDRS measures activities of daily living. Points can range from 0-52 with 0 being better outcomes and 52 being a worse outcome.
  units on a scale | 9.50 (5.40) | 11.23 (4.76) | 10.48 (5.01)
Unified Parkinson's Disease Rating Scale (UPDRS) Motor subsection (Part III) [Mean (Standard Deviation); unit: points] — This is part III of the UPDRS scale. It measures motor function in PD patients. Scores range from 0 to 108, with a score of 0 being a better outcome and 108 being a worse outcome.
  points | 12.60 (4.38) | 14.69 (5.19) | 13.78 (4.86)
Unified Parkinson's Disease Rating Scale (UPDRS) Total score [Mean (Standard Deviation); unit: units on a scale] — The UPDRS is a rating tool to follow the longitudinal course of Parkinson's Disease. It is made up of: Part 1- Mentation, Behavior, and Mood; Part 2- Activities of Daily Living (ADL); Part 3 - Motor function; and Part IV - Complications. These are evaluated by interview. Some sections require multiple grades assigned to each extremity. A total of 199 points are possible. 199 represents the worst (total disability), 0 =no disability. To get the total score you sum up each subsection score.
  units on a scale | 24.00 (9.67) | 25.08 (11.93) | 24.61 (10.78)
Parkinson's Disease Quality of Life (PDQOL) total score [Mean (Standard Deviation); unit: units on a scale] — Parkinson's disease quality of life scale has a possible point range from 37 (worst outcome) to 185 (best outcome).
  units on a scale | 124.10 (19.96) | 115.31 (10.68) | 119.13 (15.65)
Hoehn & Yahr stage [Number; unit: participants] — Stage 1: Unilateral disease. (Better outcome) Stage 1.5: Unilateral plus axial involvement. Stage 2: Bilateral disease, without impairment of balance. Stage 2.5: Mild bilateral disease, with recovery on pull test. Stage 3: Mild to moderate bilateral disease; some postural instability; physically independent. (Worst Outcome)
  participants
    Stage 1 | 1 | 0 | 1
    Stage 1.5 | 1 | 1 | 2
    Stage 2 | 1 | 2 | 3
    Stage 2.5 | 6 | 7 | 13
    Stage 3 | 1 | 3 | 4
Incontinence Quality of Life scale (IQOL) [Mean (Standard Deviation); unit: units on a scale] — The Incontinence Quality of Life scale has a possible range of 22 (worst outcome) to 110 (best outcome) total points.
  units on a scale | 78.00 (20.03) | 75.92 (18.87) | 76.83 (18.96)
Bladder diary: # micturations [Mean (Standard Deviation); unit: Micturation episodes per 24 hour period] — This is the mean number of micturations per 24 hour period as recorded on a 3-day bladder diary
  Micturation episodes per 24 hour period | 9.03 (2.21) | 9.23 (3.31) | 9.14 (2.83)
Bladder diary: # leaks [Mean (Standard Deviation); unit: Number of leaks per 24-hour period] — This is the mean number of leaks as recorded on a 3-day bladder diary.
  Number of leaks per 24-hour period | 1.33 (2.45) | 1.72 (1.23) | 1.55 (1.82)
Bladder diary: # nocturia episodes [Mean (Standard Deviation); unit: Number of nocturia episodes per 24 hours] — This is the mean number of nocturia episodes as recorded on a 3-day bladder diary.
  Number of nocturia episodes per 24 hours | 2.23 (1.69) | 1.90 (1.09) | 2.04 (1.36)
Patient perception of Bladder Condition (PBC/PPBC) [Number; unit: participants] — The PBC/PPBC is a single-item global measure for patients with overactive bladder.
  participants
    Causes me (some) moderate problems | 5 | 5 | 10
    Causes me severe problems | 4 | 7 | 11
    Causes me many severe problems | 1 | 1 | 2
Patient Perception of Intensity of Urgency Scale (PPIUS) [Number; unit: participants] — The PPIUS is a scale to assess patient's perception of their level of urgency. Mild urgency = better outcome; Severe urgency = worse outcome.
  participants
    Mild Urgency | 3 | 1 | 4
    Moderate Urgency | 4 | 5 | 9
    Moderate-Severe | 0 | 1 | 1
    Severe Urgency | 3 | 6 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Micturations Per 24 Hour Period
Description: The primary objective of this study is to measure the efficacy of solifenacin succinate (VESIcare) in reducing the mean number of micturitions per 24 hour period in Parkinson's disease (PD) patients as measured by voiding diaries.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Number of micturations per 24 hours
Arm/Group | Solifenacin Succinate (VESIcare) | Placebo
Number analyzed (Participants) | 9 | 12
Number of micturations per 24 hours
  Baseline | 8.78 (2.18) | 9.19 (3.46)
  Endpoint (12 weeks) | 8.00 (3.36) | 8.94 (3.06)
Statistical Analysis 1: Comparison: Solifenacin Succinate (VESIcare) vs Placebo; Test type: Superiority or Other; p = 0.53, ANCOVA; Adjusted for baseline value; Effect size = 0.20 — This represents the effect size between solifenacin and placebo

2. Secondary Outcome: Number of Urinary Incontinence Episodes Per 24 Hour Period
Description: This scale it the mean number of urinary incontinence episodes per 24 hour period, as assessed by a 3-day bladder diary. The goal is to examine the effect of solifenacin succinate (VESIcare) on urinary incontinence severity.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Number of incontinence episodes/24 hours
Arm/Group | Solifenacin Succinate (VESIcare) | Placebo
Number analyzed (Participants) | 9 | 12
Number of incontinence episodes/24 hours
  Baseline | 1.48 (2.56) | 1.78 (1.27)
  Endpoint (12 weeks) | 0.30 (0.31) | 1.61 (1.40)
Statistical Analysis 1: Comparison: Solifenacin Succinate (VESIcare) vs Placebo; Test type: Superiority or Other; p = 0.01, ANCOVA; Effect size = 0.53

3. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS) Total
Description: To examine the effect of solifenacin succinate (VESIcare) on Parkinson's disease severity. The UPDRS total score ranges from 0 (no disability) to 199 (total disability).
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Solifenacin Succinate (VESIcare) | Placebo
Number analyzed (Participants) | 9 | 12
units on a scale
  Baseline | 25.00 (9.70) | 25.67 (12.26)
  Endpoint (12 weeks) | 21.67 (9.59) | 25.75 (8.76)
Statistical Analysis 1: Comparison: Solifenacin Succinate (VESIcare) vs Placebo; Test type: Superiority or Other; p = 0.22, ANCOVA; Effect size = 0.35

4. Secondary Outcome: Parkinson's Disease Quality of Life Scale (PDQOL)
Description: This scale is used to assess quality of life in Parkinson's Disease patients. Parkinson's disease quality of life scale has a possible point range from 37 (worst outcome) to 185 (best outcome). The goal of this outcome measure is to examine the effect of solifenacin succinate (VESIcare) on quality of life.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Solifenacin Succinate (VESIcare) | Placebo
Number analyzed (Participants) | 9 | 12
units on a scale
  Baseline | 125.00 (20.95) | 114.50 (10.73)
  Endpoint (12 weeks) | 116.00 (26.42) | 112.92 (17.19)
Statistical Analysis 1: Comparison: Solifenacin Succinate (VESIcare) vs Placebo; Test type: Superiority or Other; p = 0.47, ANCOVA; Effect size = 0.27

5. Secondary Outcome: Number of Nocturia Episodes Per 24 Hour Period
Description: To examine the effect of solifenacin succinate (VESIcare) on urinary incontinence severity
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Number of nocturia episodes per 24 hours
Arm/Group | Solifenacin Succinate (VESIcare) | Placebo
Number analyzed (Participants) | 9 | 12
Number of nocturia episodes per 24 hours
  Baseline | 2.48 (1.59) | 1.92 (1.14)
  Endpoint (12 weeks) | 2.04 (1.96) | 1.78 (0.88)
Statistical Analysis 1: Comparison: Solifenacin Succinate (VESIcare) vs Placebo; Test type: Superiority or Other; p = 0.94, ANCOVA; Effect size = 0.11

ADVERSE EVENTS:
Arm/Group | Solifenacin Succinate (VESIcare) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/13
Other Adverse Events (participants affected / at risk) | 4/10 | 0/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Solifenacin Succinate (VESIcare) (N=10) | Placebo (N=13)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Xerostomia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No